CLINICAL TRIAL: NCT06439680
Title: The Effect of " HASCV-R" Training Program on Women's Health Promotion and Protective Behaviors: A Randomized Controlled Experimental Study
Brief Title: HASCV-R" Health Programme: a RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bozok University (Other)
Responsible Party: Principal Investigator, Mehmet KORKMAZ, Phd. Mehmet Korkmaz, Bozok University
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: 05/24
Record Dates: First submitted 2024-05-28; First posted 2024-06-03 (Actual); Last update posted 2024-06-03 (Actual); Status verified 2023-09

CONDITIONS: Health Behavior
Keywords: Health behaviors; health promotion; Women's health
MeSH Terms: conditions — Health Behavior

STUDY DESIGN:
Intervention Model Description: double-blind randomised controlled pretest-posttest experimental research
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental (Experimental): Experimental: experimental This study was carried out with the women living in Tokat province. Trainings and measurement tools in the HASCV-R programme was implemented in the Hanımeli culture and art centers.
  Interventions: Other: HASCV-R" Health Programme
- control (Other): control
  Interventions: Other: HASCV-R" Health Programme

INTERVENTIONS:
Other: HASCV-R" Health Programme — HASCV-R program "Healthy nutrition, Active life, Ways to cope with Stress, Cancer and cancer screening, Vaccination - Reproductive health" Training programme

SUMMARY:
The goal of this randomized controlled trial: is to determine the effect of " HASCV-R " health programme on the health promoting and protective behaviours of the women. The main question it aims to answer are:

• Does the HASCV-R program, positively affect the health promoting and protective behaviours of women? The health program was given to the women in the experimental group in five sessions of 40 minutes each for five weeks. The program was implemented to 45 women. After obtaining consent from women, Data were gathered with all participants at the available time and places.

The data were collected from the control and experimental groups at two different times, prior to the program was implemented and 3 months after the program was implemented.

DETAILED DESCRIPTION:
Positive health behaviors aimed at improving health refer to individuals' conscious efforts to protect and improve their own health and the health of other individuals. Examples of positive health behaviors include eating adequate and balanced nutrition, paying attention to sleep patterns, doing physical activity, staying away from stress, having regular health checks, and communicating effectively and positively with people. In order for individuals to acquire positive health behaviors, they need to have an idea about all of these behaviors and turn the knowledge they have acquired into behavior. Health professionals undoubtedly have a large share in the formation of this health awareness, as well as in the treatment of diseases, as well as in protecting health and avoiding risky health behaviors.

It is seen that in developed societies, the planning, implementation and evaluation stages of health promotion programs in health services are carried out by professional nurses. The group that will ensure the development of health, informing and guiding healthy behaviors are nurses who provide professional care in health institutions. There are training programs to improve women's health in the literature, but there is no training program that is both health-promoting and health-protective. Considering the impact of nurses on health education and creating behavioral change, their knowledge on this subject and their ability to transfer this to public health is of great importance. In addition, considering that a healthy lifestyle has become so important today, the unique value of the study is that the training program to be developed includes behaviors that promote and protect women's health. This research was planned to evaluate the effect of the "HASCV-R" training program on women's health-promoting and protective behaviors.

ELIGIBILITY:
Inclusion Criteria:

* volunteering to participate in the study,
* be between the ages of 18 and 49,
* being a women,
* no communication barriers (to communicate with any problem such as hearing problem, speech impediment),
* to be married

Exclusion Criteria:

being younger than 18 or over 49,

* be man,
* ınability to communicate with any problem such as hearing problem, speech impediment,
* living single,
* refusing to participate in the study

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 90 (Actual)
Dates: Start 2023-05-15 (Actual); Primary Completion 2023-09-15 (Actual); Study Completion 2023-11-15 (Actual)

PRIMARY OUTCOMES:
Questionnaire form | prior to the program was implemented and 3 months after the program was implemented
  This form, developed by the researchers based on the literature, includes the socio-demographic characteristics of the women such as age, education status, income status, etc.)

SECONDARY OUTCOMES:
Health Promoting and Protective Behaviours Scale | prior to the program was implemented and 3 months after the program was implemented
  Evaluates the extent to which the individual keeps himself active in daily life, regular exercise behaviours and behaviours related to meeting physiological needs such as eating and drinking.
Scale for Determining Reproductive Health Protective Attitudes of Married Women | prior to the program was implemented and 3 months after the program was implemented
  It was developed to determine the reproductive health protective attitudes and behaviours of married women.

CONTACTS AND LOCATIONS:
Locations (1):
- Yozgat Bozok University, Yozgat, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No